CLINICAL TRIAL: NCT01736319
Title: Artemisinin-resistant Plasmodium Falciparum Malaria in Cambodia
Brief Title: Artemisinin-resistant Malaria in Cambodia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912163; 12-I-N163
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2016-04-06

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Artemisinin-based Combination Therapies; Recrudescence; DHA-PPQ; Parasite Clearance Rate
MeSH Terms: conditions — Malaria, Falciparum; Recurrence

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Artemisinin-based combination therapies (ACTs) are the first-line treatments for malaria. ACTs are highly effective, but malaria caused by the Plasmodium falciparum parasite is becoming resistant to some ACTs. ACT-resistant malaria has shown up in some parts of Cambodia, but not yet in other parts of the country. This has been shown by treating patients with ACTs, checking the amount of parasites in the patient s blood every 6 hours, and calculating the rate of parasite clearance. The parasite clearance rate in response to ACTs is getting slower in western Cambodia and may be the first sign of ACT resistance. Researchers want to study how effective ACTs are in different regions of Cambodia. This study will look at the extent of ACT resistance and how widespread ACT-resistant malaria has become.

Objectives:

- To compare the prevalence of ACT-resistant malaria in western, northern and eastern Cambodia.

Eligibility:

- Individuals between 2 and 65 years of age who have uncomplicated Plasmodium falciparum malaria and have not taken any antimalarial drugs for their symptoms in the previous 7 days.

Design:

* Participants will be recruited from clinics and hospitals in three Cambodian provinces.
* Participants will be informed about the study and their consent to participate in the study will be obtained.
* A venous blood sample will be obtained from patients before treatment and used for laboratory experiments to measure parasite and patient factors that might affect the parasite clearance rate.
* Participants with malaria will be treated with dihydroartemisinin-piperaquine (DHA-PPQ), the standard first-line treatment for malaria in Cambodia.
* Treatment will be monitored with frequent blood samples obtained from a finger prick. The amount of malaria parasites in each blood sample will be counted and followed until they are no longer detectable.
* Participants will have weekly follow-up visits for up to 9 weeks. Finger-prick blood samples will be taken at each visit to see if the parasites reappear after treatment with ACT.

DETAILED DESCRIPTION:
Artemisinin-based combination therapies (ACTs) are the first-line treatments for Plasmodium falciparum malaria worldwide. In Western Cambodia,artemisinin resistance has been defined as a long half-life of parasite clearance (T1/2) in response to an artemisinin, given orally for uncomplicated malaria. We hypothesize that this artemisinin resistance phenotype compromises the efficacy of ACTs. The primary objective of this study is to compare P. falciparum recrudescence rates in Western, Northern and Eastern Cambodia, following dihydroartemisinin-piperaquine (DHA-PPQ) treatment. The secondary objective of this study is to determine whether parasite recrudescence is associated with long T1/2. In the Parasite Recrudescence Study, patients with uncomplicated malaria will receive directly-observed treatment with DHA-PPQ over 3 days. We will follow these patients weekly for 9 weeks to identify those with recurrent parasitemia and use genotyping methods to distinguish recrudescences from reinfections. We will enroll a subset of these patients who have an initial parasite density greater than or equal to 10,000/microL in the Parasite Clearance Rate Study and follow their parasite densities more intensively by examining 6-hourly finger prick blood samples until parasites are undetectable by microscopy. With these data we will calculate and compare T1/2 values from patients with and without recrudescent parasitemia. Using various laboratory assays, we will also explore the contribution of host factors to T1/2 variation, and whether naturally-acquired immunity reduces the risk of drug-resistant parasite recrudescence.

ELIGIBILITY:
* INCLUSION CRITERIA (Parasite Recrudescence Study):

  1. Age 2 to 65 years, inclusive
  2. Uncomplicated P. falciparum malaria
  3. Temperature greater than or equal to 37.5 degrees Celsius or history of fever within the last 24 h
  4. P. falciparum asexual parasite density less than or equal to 200,000/microL
  5. Willingness to allow the storage of blood samples collected as part of the study
  6. Willingness and ability of patients/guardians to comply with the protocol for the duration of the study.

EXCLUSION CRITERIA (Parasite Recrudescence Study):

1. Severe malaria: diminished consciousness, respiratory distress, severe prostration, anuria, jaundice, hemoglobinuria, repetitive vomiting, or cessation of eating and drinking
2. Non-malaria etiology of febrile illness (e.g., respiratory tract infection) evident by history and physical examination
3. Hematocrit <25%
4. Treatment of present symptoms with an antimalarial drug within the previous 7 days
5. Pregnancy or breastfeeding
6. History of allergy or known contraindication to artemisinins or MQ
7. Splenectomy
8. P. vivax parasitemia

INCLUSION CRITERIA (Peripheral Blood Collection Study):

1. Healthy-appearing adults greater than or equal to 18 years old
2. Residence in Pursat province
3. Willingness to participate in the study as evidenced by informed consent

EXCLUSION CRITERIA (Peripheral Blood Collection Study):

1. Pregnancy
2. Hematocrit <25%

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2012-06-26; Study Completion 2016-04-06

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Center for Parasitology, Entomology, and Malaria Controk, Ministry of H, Phnom Penh, Cambodia

REFERENCES:
- [Background] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202
- [Background] Phyo AP, Nkhoma S, Stepniewska K, Ashley EA, Nair S, McGready R, ler Moo C, Al-Saai S, Dondorp AM, Lwin KM, Singhasivanon P, Day NP, White NJ, Anderson TJ, Nosten F. Emergence of artemisinin-resistant malaria on the western border of Thailand: a longitudinal study. Lancet. 2012 May 26;379(9830):1960-6. doi: 10.1016/S0140-6736(12)60484-X. Epub 2012 Apr 5. PMID 22484134
- [Background] White NJ. The parasite clearance curve. Malar J. 2011 Sep 22;10:278. doi: 10.1186/1475-2875-10-278. PMID 21939506
- [Derived] Amaratunga C, Lim P, Suon S, Sreng S, Mao S, Sopha C, Sam B, Dek D, Try V, Amato R, Blessborn D, Song L, Tullo GS, Fay MP, Anderson JM, Tarning J, Fairhurst RM. Dihydroartemisinin-piperaquine resistance in Plasmodium falciparum malaria in Cambodia: a multisite prospective cohort study. Lancet Infect Dis. 2016 Mar;16(3):357-65. doi: 10.1016/S1473-3099(15)00487-9. Epub 2016 Jan 8. PMID 26774243
- [Derived] Witkowski B, Amaratunga C, Khim N, Sreng S, Chim P, Kim S, Lim P, Mao S, Sopha C, Sam B, Anderson JM, Duong S, Chuor CM, Taylor WR, Suon S, Mercereau-Puijalon O, Fairhurst RM, Menard D. Novel phenotypic assays for the detection of artemisinin-resistant Plasmodium falciparum malaria in Cambodia: in-vitro and ex-vivo drug-response studies. Lancet Infect Dis. 2013 Dec;13(12):1043-9. doi: 10.1016/S1473-3099(13)70252-4. Epub 2013 Sep 11. PMID 24035558